CLINICAL TRIAL: NCT03006393
Title: Dynamics of Inflammation and Its Blockade on Motivational Circuitry in Depression
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Michael Treadway, Assistant Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB00087941; R01MH108605 (NIH)
Record Dates: First submitted 2016-12-28; First posted 2016-12-30 (Estimated); Results first posted 2021-10-19 (Actual); Last update posted 2021-11-18 (Actual); Status verified 2021-10

CONDITIONS: Depression
Keywords: Neuroscience; Behavioral; Social
MeSH Terms: conditions — Depression; Behavior | interventions — Infliximab; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Infliximab (Experimental): Participants randomized to the infliximab group will receive one infusion of infliximab at 5mg/kg body weight.
  Interventions: Drug: Infliximab
- Placebo (Placebo Comparator): Participants randomized to the placebo group will receive one placebo infusion.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Infliximab — One infusion of Infliximab (Remicade) will be administered intravenously (IV) at 5 mg/kg body weight over a two hour period.
  Other Names: Remicade
  Arms: Infliximab
Other: Placebo — One infusion of placebo treatment will be administered intravenously (IV) over a two hour period.
  Other Names: Saline Solution
  Arms: Placebo

SUMMARY:
The main purpose of this study is to examine the effects of infliximab on measures related to depression symptoms. Infliximab is also known by its brand name Remicade. Infliximab, or Remicade, is given to by an intravenous (IV) needle and is currently used to treat rheumatoid arthritis and Crohn's disease. Infliximab is thought to help these conditions because it reduces inflammation in the body. Infliximab (Remicade) reduces inflammation by blocking a chemical in the body called tumor necrosis factor (TNF)-alpha. This chemical produces inflammation. Inflammatory chemicals in the body like TNF-alpha appear to be increased in some people with major depression. Researchers believe that a drug like infliximab, which blocks TNF-alpha, may be helpful in treating depression.

This is a double-blind, placebo-controlled study in which participants will be randomized to receive one infusion of infliximab or placebo. The study will assess neuroimaging measures of corticostriatal circuitry before and after a placebo-controlled pharmacologic blockade of inflammation in 80 depressed patients.

DETAILED DESCRIPTION:
The main purpose of this study is to examine the effects of infliximab on measures related to depression symptoms. Infliximab is also known by its brand name Remicade. Infliximab, or Remicade, is given by an intravenous (IV) needle and is currently used to treat rheumatoid arthritis and Crohn's disease. Infliximab is thought to help these conditions because it reduces inflammation in the body. Infliximab (Remicade) reduces inflammation by blocking a chemical in the body called tumor necrosis factor (TNF)-alpha. This chemical produces inflammation. Inflammatory chemicals in the body like TNF-alpha appear to be increased in some people with major depression. Researchers believe that a drug like infliximab, which blocks TNF-alpha, may be helpful in treating depression.

This is a double-blind, placebo-controlled study in which participants will be randomized to receive one infusion of infliximab or placebo. This study will assess neuroimaging measures of corticostriatal circuitry before and after a placebo-controlled pharmacologic blockade of inflammation in 80 depressed patients (n = 40 per group) recruited to ensure high levels of peripheral inflammation (CRP > 3mg/L).

Primary aims are to evaluate whether 1) corticostriatal function during reward motivation and anticipation are associated with change in peripheral inflammation following pharmacologic blockade relative to placebo 2) the temporal dynamics of change in inflammation, gene- expression, reward motivation and reinforcement learning behavior and motivational symptoms assessed at baseline, and 24 hours, 3 days, 1 week and two weeks post infliximab infusion, and 3) test an integrative multi- level path model to determine whether change in corticostriatal circuitry following inflammation blockade mediates the relationship between change in inflammation and change in motivational anhedonia symptoms.

These data will provide further validation of inflammatory cytokines as therapeutic targets for motivational symptoms in depression and will define symptom targets and biomarkers of response for future studies.

ELIGIBILITY:
Inclusion Criteria:

* All subjects will be fully ambulatory and in good medical health. Note: By Diagnostic and Statistical Manual of Mental Disorders (DSM-4) definition of depression, subjects will report impairment in ability to carry out daily activities as a result of their major depression.
* Subjects will be able to read and understand English.
* Women must be postmenopausal (no menstrual period for a minimum of 1 year) or surgically sterilized and/or have a negative serum pregnancy test within thirty days of infusion (may be repeated closer to infusion date if deemed necessary by the PI or PI's designee) and negative urine pregnancy tests throughout the study (performed at each visit after the serum pregnancy test is completed).
* Men and women of childbearing potential must use adequate birth control measures (e.g., abstinence, oral contraceptives, intrauterine device, barrier method with spermicide, implantable or injectable contraceptives or surgical sterilization) for the duration of the study and should continue such precautions for 6 months after receiving the last infusion.

The following are considered eligible according to the following tuberculosis (TB) screening criteria:

* Have no history of latent or active TB prior to screening.
* Have no signs or symptoms suggestive of active TB upon medical history and/or physical examination.
* Have had no recent close contact with a person with active TB or, if there has been such contact, will be referred to a physician specializing in TB to undergo additional evaluation to rule out infection. The candidate will be excluded from study participation if the specialist diagnoses active TB and or determines TB treatment is warranted.
* Have a chest radiograph (both posterior-anterior and lateral views), taken within 3 months prior to the first administration of study agent and read by a qualified radiologist, with no evidence of current active TB or old inactive TB.
* History of negative purified protein derivative (PPD) test; or documentation of a negative blood test (Quantiferon-TB-Gold). Any candidate testing positive for tuberculosis in the medical screening evaluation, will be excluded from study participation

Exclusion Criteria:

* Subjects will be excluded for any prior use of a TNF-alpha antagonist (i.e. etanercept, infliximab, adalimumab) and/or use of any other immunosuppressant agent (i.e. systemic corticosteroids or anti-proliferative agents such as methotrexate) within one year of study entry.
* Subjects chronically (i.e. more than one month) taking more than the equivalent of 2 mg of lorazepam a day of a benzodiazepine will be excluded.
* Subjects will be required not to use anti-inflammatory agents, non-steroidal anti-inflammatory agents (NSAIDs) (excluding 81mg of aspirin), glucocorticoid containing medicines or statins, or cyclooxygenase-2 (COX-2) inhibitors during the study as these agents may interfere with assessment of the relationship between inflammatory markers and treatment response.

Note: Acetaminophen will be allowed.

Potential subjects will be excluded for a history of any of the following conditions:

* Abnormal electrocardiogram
* Auto-immune condition as confirmed by laboratory testing (i.e. rheumatoid arthritis, inflammatory bowel disease, multiple sclerosis, lupus)
* History of significant infectious sequelae, including but not limited to, abscess or sepsis
* Infection within one month prior to screening that required antibiotic or antiviral therapy
* History of a more than mild cognitive disorder or ≤ 24 on the Mini-Mental State Exam (MMSE), unless otherwise approved by PI or his designee
* Unstable cardiovascular or endocrinologic disease (as determined by physical examination and/or laboratory testing)
* Any other current or past medical condition that might increase the risk of infliximab-related adverse events
* Potential subjects will be excluded for any of the following conditions:
* Active suicidal ideation defined as a score of ≥3 on Columbia Suicide Severity Rating Scale (C-SSR).
* Suicide attempt within six months of study entry
* Schizophrenia or Schizoaffective Disorder
* Active Eating Disorder (excluding binge-eating disorder)
* History of any (non-mood related) psychotic disorder or active psychotic symptoms of any type

Subjects will have had no infectious illnesses for one month prior to infusion. Should a subject develop an infection (i.e. flu, upper respiratory viral infection) between screening and infusion, the infusion will be delayed until 4 weeks after resolution of symptoms. As noted above, patients with a chronic infectious condition or with a past history of serious infectious complications will be excluded.

Subjects will be excluded for any evidence on laboratory testing (or by history) of hematologic, renal or hepatic abnormality. Subjects will be excluded for a positive anti-nuclear antibody (ANA) test.

Infliximab Related Exclusion Criteria:

* Have had any previous treatment with monoclonal antibodies or antibody fragments.
* History of receiving human/murine recombinant products or a known allergy to murine products. A known allergy to murine product is definitely an exclusion criterion.
* Documentation of seropositive for human immunodeficiency virus (HIV). Any candidate testing positive for HIV, in the medical screening evaluation, will be excluded from study participation.
* Documentation of a positive test for hepatitis B surface antigen or hepatitis C. Any candidate testing positive for hepatitis B or hepatitis C, in the medical screening evaluation, will be excluded from study participation.
* Are unable or unwilling to undergo multiple venipunctures because of poor tolerability or lack of easy access.
* Use of any investigational drug within 30 days prior to screening or within 5 half-lives of the investigational agent, whichever is longer.
* Presence of a transplanted solid organ (with the exception of a corneal transplant > 3 months prior to screening).
* Have a concomitant diagnosis or history of congestive heart failure.
* Have a history of alcohol or substance abuse within the preceding 6 months that, in the opinion of the investigator, may increase the risks associated with study participation or study agent administration, or may interfere with interpretation of results. (As determined by Structured Clinical Interview for DSM-5 (SCID-5))
* Have a known history of serious infections (e.g., hepatitis, pneumonia, or pyelonephritis) in the previous 3 months.
* Have or have had an opportunistic infection (e.g., herpes zoster [shingles], cytomegalovirus, Pneumocystis carinii, aspergillosis, histoplasmosis, or mycobacteria other than TB) within 6 months prior to screening.
* Have a history of lymphoproliferative disease, including lymphoma or signs suggestive of possible lymphoproliferative disease such as lymphadenopathy of unusual size or location (e.g., nodes in the posterior triangle of the neck, infraclavicular, epitrochlear, or periaortic area), or splenomegaly.
* Currently have any known malignancy other than the condition being treated or have a history of malignancy within the previous 5 years, with the exception of basal cell or squamous cell carcinoma of the skin that has been fully excised with no evidence of recurrence.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2020-09-26 (Actual); Study Completion 2020-09-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Treadway, PhD, Principal Investigator — Emory University
Locations (1):
- Emory University, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lee Y, Subramaniapillai M, Brietzke E, Mansur RB, Ho RC, Yim SJ, McIntyre RS. Anti-cytokine agents for anhedonia: targeting inflammation and the immune system to treat dimensional disturbances in depression. Ther Adv Psychopharmacol. 2018 Nov 19;8(12):337-348. doi: 10.1177/2045125318791944. eCollection 2018 Dec. PMID 30524702

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at Emory University in Atlanta, Georgia, USA. Enrollment began in August 2016 and all follow up was complete by September 26, 2020.
Groups:
- Infliximab: Participants randomized to the infliximab group received one infusion of Infliximab (Remicade) administered intravenously (IV) at 5 mg/kg body weight over a two hour period.
- Placebo: Participants randomized to the placebo group received one infusion of placebo treatment administered intravenously (IV) over a two hour period.
Period: Overall Study
Arm/Group | Infliximab | Placebo
Started | 21 | 21
Completed | 20 | 18
Not Completed | 1 | 3
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Pregnancy | 0 | 1
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Infliximab | Placebo | Total
Number analyzed (Participants) | 21 | 21 | 42
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.1 (9.2) | 38.0 (7.9) | 39.03 (8.53)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 19 | 37
  Male | 3 | 2 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 2 | 5
  Not Hispanic or Latino | 18 | 18 | 36
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 3 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 8 | 12 | 20
  White | 13 | 5 | 18
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 21 | 21 | 42

OUTCOME MEASURES:

1. Primary Outcome: Effort-based Decision-making (EBDM) Task Score
Description: Reward motivation was assessed by a laboratory effort-based decision-making (EBDM) task. On each trial, participants make a choice about expending more or less physical effort (rapid button pressing) in exchange for varying amounts of monetary rewards. Models of subjective value were fit to each participants' data using maximum likelihood estimation and were compared using Bayesian Information Criterion to identify the model that provides the best fit for participants' responses. Discounting functions were based on previous work and include linear, quadratic, hyperbolic, flexible power models. Models considering the potential effects of fatigue and examination of post-scan switching behavior were also evaluated. The best-fitting model from baseline data was applied to look at changes related to infliximab. Reported values reflect a model-derived summary statistic for effort discounting behavior, without a fixed range, where lower values associated with greater motivation.
Time Frame: Baseline, Day 14
Population: This analysis includes participants who completed the indicated study visit.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Infliximab | Placebo
Number analyzed (Participants) | 21 | 21
score on a scale
  Baseline | 2.13 (1.76) | 2.09 (1.52)
  Day 14: number analyzed (Participants) | 20 | 18
  Day 14 | 1.85 (1.28) | 2.78 (1.70)

2. Secondary Outcome: Plasma C-reactive Protein (CRP) Level
Description: C-reactive protein (CRP) is a blood test marker for inflammation in the body. CRP is produced in the liver and its level is measured by testing the blood. CRP level was measured at baseline and Day 14. Lower result correlates with better outcome.
Time Frame: Baseline, Day 14
Population: This analysis includes participants who completed the indicated study visit and had usable blood samples. Some participants did not complete the trial and another participant had a blood sample of poor quality.
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Infliximab | Placebo
Number analyzed (Participants) | 20 | 21
mg/L
  Baseline | 4.18 (3.28) | 7.81 (7.85)
  Day 14: number analyzed (Participants) | 19 | 18
  Day 14 | 2.78 (4.63) | 6.35 (6.96)

3. Secondary Outcome: Plasma Interleukin-6 (IL-6) Level
Description: Plasma IL-6 level will be collected via blood draw. IL-6 level was collected at baseline and Day 14. Lower result correlates with better outcome.
Time Frame: Baseline, Day 14
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Infliximab | Placebo
Number analyzed (Participants) | 20 | 21
pg/ml
  Baseline | 1.13 (0.96) | 1.07 (0.97)
  Day 14: number analyzed (Participants) | 19 | 18
  Day 14 | 0.97 (1.00) | 1.19 (1.25)

ADVERSE EVENTS:
Time Frame: Adverse events were tracked from the time of consent through the 30-Day Post-Infusion Follow-Up Phone Call.
Arm/Group | Infliximab | Placebo
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/21
Other Adverse Events (participants affected / at risk) | 19/21 | 13/21
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Infliximab (N=21) | Placebo (N=21)
Headache (General disorders) | 8 (8) | 8 (8)
Heartburn (Gastrointestinal disorders) | 2 (2) | 0 (0)
Menstruation (Reproductive system and breast disorders) | 1 (1) | 2 (2)
Bruises (Vascular disorders) | 5 (5) | 5 (5)
Syncope (General disorders) | 1 (1) | 0 (0)
Pain in joints (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Sore throat (General disorders) | 4 (4) | 0 (0)
Bloody stool (Gastrointestinal disorders) | 1 (1) | 1 (1)
Pain in leg (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Chills (General disorders) | 0 (0) | 1 (1)
Allergies (General disorders) | 1 (1) | 2 (2)
Dizziness (General disorders) | 2 (2) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2) | 1 (1)
Chest pain (General disorders) | 1 (1) | 0 (0)
Change in urination (Renal and urinary disorders) | 2 (2) | 0 (0)
Change in blood pressure (General disorders) | 1 (1) | 0 (0)
Muscle tension (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Itchiness (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2)
Motor vehicle accident (General disorders) | 1 (1) | 1 (1)
Pain in neck (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Stomach ache (Gastrointestinal disorders) | 1 (1) | 1 (1)
Numbness (Nervous system disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 2 (2) | 0 (0)
Migraine (Nervous system disorders) | 1 (1) | 0 (0)
Swelling (General disorders) | 1 (1) | 2 (2)
Laceration (Musculoskeletal and connective tissue disorders) | 11 | 0 (0)
Change in appetite (General disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-07-06): https://cdn.clinicaltrials.gov/large-docs/93/NCT03006393/Prot_SAP_000.pdf
  • Informed Consent Form (2019-11-26): https://cdn.clinicaltrials.gov/large-docs/93/NCT03006393/ICF_001.pdf